CLINICAL TRIAL: NCT06824532
Title: Veteran's Perceptions of Ketamine-Assisted Psychotherapy (KAP) for Depression and End-of-Life
Brief Title: Veteran's Perceptions of Ketamine-Assisted Psychotherapy for Depression and End-of-Life
Acronym: KAP
Status: Recruiting | Type: Observational
Sponsor: Albany Research Institute, Inc. (Other)
Responsible Party: Principal Investigator, Caitlin Holley, Psychologist, Albany Research Institute, Inc.
Other Study IDs: AlbanyRI
Record Dates: First submitted 2025-02-06; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this exploratory, mixed-method design study is to gather qualitative and quantitative data obtained through interviews and questionnaires with veterans who are currently enrolled at the VA for healthcare. The main question this study aims to answer is: How do veterans aged 65+ who are enrolled for care at the VA understand ketamine assisted psychotherapy for depression and for end-of-life distress? Using a story-completion approach, participants will be provided with a brief story starter involving a fictitious character and scenario and asking them to complete the story. Few contextual details will be offered about the character. In responding to ambiguous cues, participants are thought to project their conscious and subconscious perceptions about the phenomenon in question onto the story, a useful method for exploring stigmatized topics. The purpose of this exercise is to ascertain the participants attitudes and perceptions regarding ketamine assisted psychotherapy.

DETAILED DESCRIPTION:
Veterans will be informed of the study by their VA providers (Behavioral Health Clinic, Primary Care, etc). Veterans who are interested will have their contact information passed on to the study investigators. Once screened and enrolled in the study veterans will complete a brief demographics form, and three brief symptom screening questionnaires: Patient Health Questionnaire 9, Ten Item Personality Inventory, and the Death Anxiety Questionnaire. Participants then engage in the recorded interview during which they are provided with a brief story starter, as described above. In the story, a fictitious veteran with a diagnosis of depression is offered an opportunity to engage in ketamine assisted psychotherapy (KAP). The veteran then receives a cancer diagnosis and is again offered a chance to consider KAP. Participants are asked to share what questions, concerns, hopes, and expectations may be present for the fictitious veteran in the story. Interviews will then be transcribed and the PI and the collaborators will read all transcriptions and generate recurring themes that can be reliably coded. The investigators will then code the transcripts for the presence of themes. Data analytic plans include calculating the prevalence of each theme and examining their correlates with measures of severity of symptoms as well as any demographic variables. It is hoped that this data can inform educational and other roll-out efforts within the VA system around KAP.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled in VA care.
* Age 65 or older.
* Fluent in written and spoken English.

Exclusion Criteria:

* Cognitively impaired to the extent that patient cannot comprehend the survey.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The demographic makeup of the sample mimics the demographic makeup of the population of veterans served by VA. As such, the racial distributions will likely be primarily Caucasian, the sample is likely to be predominantly male, ranging in age from 20-100, with an average of 58 years.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 | 2 weeks
  Screening tool for depressive symptoms. Scores range from 0-27 with lower scores indicating better outcomes
Ten Item Personality Inventory | 2 weeks
  A 10-item measure of the Big Five dimensions is offered for situations when very short measures are needed, personality is not the primary topic of interest. It assesses the big-five traits-Emotional Stability, Extraversion, Openness, Agreeableness, and Conscientiousness-using two items for each scale. Scores range from 1-70.
Death Anxiety Questionnaire | 2 weeks
  The 15-item self report scale is a reliable and valid measure of individual differences in and perceptions of death anxiety. Scores range from 0-30 with higher scores indicate a higher level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Holley, Ph.D., Principal Investigator — Albany Research Institute, Inc.
Locations (1):
- Stratton VA Medical Center, Albany, New York, United States